CLINICAL TRIAL: NCT01658774
Title: Impact of Repeated Anthelminthic Treatment on Malaria in School Children: an Individual Randomized, Double-blind, Placebo-controlled Trial in Western Kenya
Brief Title: Impact of Repeated Anthelmintic Treatment on the Risk of Malaria in Kenyan School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: European Union (Other); Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2242; 241642 (Other Grant/Funding Number: European Union)
Record Dates: First submitted 2012-07-19; First posted 2012-08-07 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2014-02

CONDITIONS: Intestinal Helminthiasis; Ascariasis; Hookworm; Malaria
MeSH Terms: conditions — Intestinal helminthiasis; Ascariasis; Ancylostomiasis; Malaria | interventions — Albendazole; Ascorbic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Albendazole & Vitamin C (Active Comparator): Anthelmintics. A single dose of Albendazole (400mg) at month 0 and single dose of Vitamin C (500 mg) at 3, 6, 9 and 12 months.
  Interventions: Drug: Albendazole; Dietary Supplement: Vitamin C
- Albendazole (Experimental): Anthelmintics. A single does of Albendazole (400mg) every three months for 12 months
  Interventions: Drug: Albendazole

INTERVENTIONS:
Drug: Albendazole — Single 400mg dose
  Other Names: Zentel
Dietary Supplement: Vitamin C — 500 mg Vitamin C
  Arms: Albendazole & Vitamin C

SUMMARY:
Many school children in Kenya are infected with plasmodia and helminth species and are at risk of coinfection. It has been suggested that the immune response evoked by helminth infections may modify immune responses to plasmodia species and consequently alter infection and disease risks. However, studies conducted to date have been typically cross-sectional and produced conflicting results, and there is a need for longitudinal studies to better understand the clinical consequences for individuals harbouring coinfection. This study aims to investigate the impact of intensive (once every 3 months) anthelminthic treatment versus annual treatment on the risk of clinical malaria and on immune responses among school children aged 5-14 years in Western Province. Specifically, this study aims to investigate the impact of intensive anthelminthic treatment on (i) the incidence of clinical malaria in school children, assessed using active case detection; (ii) the prevalence and density of Plasmodium spp. infection, using repeat cross-sectional surveys; and (iii) malaria and helminth specific immune responses. The study hypothesis is that intensive anthelminthic treatment among children infected with either Ascaris lumbricoides or hookworm modifies human host immune responses to plasmodia and helminth infections, and therefore alters the risk of Plasmodium infection and clinical disease.

This individually randomised trial will recruit 1,450 children aged 5-14 years found to be infected with either Ascaris lumbricoides or hookworm species. Recruited children will be randomized to receive albendazole treatment either every three months or annually and monitored through periodic surveillance for clinical malaria episodes over 18 months. In addition, blood samples will be collected from sub-sample of children and screened for malaria specific immunoglobulin (Ig)G1 and IgG3 and helminth specific IgE, IgG2, IgG4 and IgM. Cell culture supernatants will be assayed for interferon (IFN)-γ, tumor necrosis factor (TNF)-α, interleukin (IL)-10, IL-5, IL-4 and IL-2.

DETAILED DESCRIPTION:
This will be an individual randomized, single-blind trial to evaluate the impact of intensive versus annual anthelminthic treatment on the incidence of clinical malaria in healthy school children.

The target population includes children attending primary school in western Kenya. The accessible population includes children attending the participating primary schools in standards 1-7 in western Kenya. The unit of analysis is the individual child. Children with informed consent and assent will be screened for helminth infections and those children found to be infected with either Ascaris lumbricoides or hookworm species will be recruited into the study. These children will be randomized to one or two groups, receiving either albendazole treatment every three months or albendazole at the start of the study and placebo every three months thereafter. Cross-sectional health surveys will be conducted before the intervention and at 6, 12 and 18 months follow-up. Weekly active case detection during school visits will be undertaken.

ELIGIBILITY:
Inclusion Criteria:

* Pupils enrolled at participating schools in classes 1-7.
* Provision of informed consent from parent or legal guardian.
* Provision of assent by student.
* Detectable infection with A.lumbricoides, T. trichiura and/or hookworm species.

Exclusion Criteria:

* Pupils unwilling to participate in the study.
* Pupils who are infected with S. haematobium or S. mansoni. These children will be treated with praziquantel.
* Known or suspected sickle-cell trait.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2377 (Actual)
Dates: Start 2013-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Incidence of clinical malaria | 18 months
  Incidence of clinical malaria, defined as fever (axillary temperature > 37.5 °C) or a reported history of fever within the preceding 24 hours in conjunction with a slide positive for Plasmodium spp. parasites at any density during 18 months of follow-up.

SECONDARY OUTCOMES:
Prevalence and density of Plasmodium spp. infection. | 18 months
Antibody isotype response to Plasmodium antigens. | 18 months
  ELISA analysis will be carried out to determine IgG1and IgG3 antibody response to Plasmodium antigens (schizont extract and Merozoite Surface Proteins (MSP)
Antibody isotype response to helminth antigens. | 18 months
  ELISA analysis will be carried out to determine and IgE, IgG2, IgG4 and IgM responses to hookworm and Ascaris lumbricoides.

CONTACTS AND LOCATIONS:
Overall Officials: Simon J Brooker, DPhil, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- KEMRI-Wellcome Trust Programme, Nairobi, Kenya

REFERENCES:
- [Derived] Kepha S, Nuwaha F, Nikolay B, Gichuki P, Mwandawiro CS, Mwinzi PN, Odiere MR, Edwards T, Allen E, Brooker SJ. Effect of Repeated Anthelminthic Treatment on Malaria in School Children in Kenya: A Randomized, Open-Label, Equivalence Trial. J Infect Dis. 2016 Jan 15;213(2):266-75. doi: 10.1093/infdis/jiv382. Epub 2015 Jul 13. PMID 26170395
- See also: Training Health Researchers into Vocational Excellence in East Africa — http://thrive.or.ug/